CLINICAL TRIAL: NCT04016402
Title: Targeting Functional Improvement in rTMS Therapy
Brief Title: Imaging to Improve Brain Stimulation
Status: Active, not recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency); Brown University (Other)
Responsible Party: Sponsor
Other Study IDs: D3152-R-1; N2864-C (Other Grant/Funding Number: Center for Neurorestoration and Neurotechnology)
Record Dates: First submitted 2019-06-19; First posted 2019-07-11 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Depressive Disorder
Keywords: Transcranial Magnetic Stimulation; Magnetic Resonance Imaging
MeSH Terms: conditions — Depressive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — None Retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study Group: All participants enrolled in the study
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Clinical transcranial magnetic stimulation administered as part of usual care for the study population
  Other Names: transcranial magnetic stimulation, theta burst transcranial magnetic stimulation

SUMMARY:
This study investigates how brains change as a result of a treatment for depression called repetitive transcranial magnetic stimulation (rTMS). People who receive rTMS will have pictures of their brains and brain activity taken by a magnetic resonance imaging (MRI) scanner before and after their treatment, as well as up to three times during the six-week treatment course. These images will be examined to see if the rTMS is placed correctly to help treat their symptoms, and what changes in brain activity are happening during the rTMS treatment

DETAILED DESCRIPTION:
Veteran patients can be referred to receive a Neuromodulation Clinic consult at the Providence VA Medical Center (PVAMC). Following this consultation, patients who are to begin rTMS therapy for the treatment of major depressive disorder (MDD) will be recruited to participate in this study. About 1 week prior to the scheduled beginning of rTMS therapy, research participants who provide informed consent will complete baseline neuropsychological measures. Within a few days of completing these measures, and before beginning rTMS therapy, participants will receive an MRI scan, including structural and functional imaging. Participants will have a similar set of MRI scans up to three times during the course of rTMS therapy, and complete neuropsychological measures at these scanning sessions. A final MRI scan will be conducted within a week of completing the rTMS therapy course, and neuropsychological measures will be completed at this session.

ELIGIBILITY:
Inclusion Criteria:

* Veteran beginning TMS therapy for the treatment of MDD at the Providence VAMC Neuromodulation Clinic
* Age between 18 and 80 years
* Able to read, verbalize, understand, and voluntarily sign the informed consent form
* Structured Clinical Interview for DSM-5 (SCID-5) confirmed diagnosis of MDD

Exclusion Criteria:

* Contraindications to MRI (e.g. implanted metal or electronic devices)
* Montreal Cognitive Assessment (MoCA) score < 26
* Pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans who receive TMS therapy for the treatment of MDD at the Providence VAMC Neuromodulation Clinic
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Distance between treatment location and brain target | Within one week of the conclusion of clinical rTMS therapy course
  A marker visible on MRI will be placed on the treatment location for the MRI scan after treatment completion. Functional MRI will be used to localize the dorsolateral prefrontal cortex (DLPFC), the brain region targeted by rTMS. The distance between these two points will be calculated for each participant.

SECONDARY OUTCOMES:
World Health Organization Disability Assessment Schedule 2.0 36-item version | Within one week before beginning clinical rTMS therapy course, 3 times during the clinical rTMS therapy course (typically 6 weeks), and within one week after the conclusion of clinical rTMS therapy course
  Scores from the World Health Organization Disability Assessment Schedule 36-item version (WHODAS-36). Self-assessment of global functioning, with scores ranging from 0 (no disability) to 100 (full disability).
Inventory of Depressive Symptoms Self-Report | Within one week before beginning clinical rTMS therapy course, 3 times during the clinical rTMS therapy course (typically 6 weeks), and within one week after the conclusion of clinical rTMS therapy course
  Scores from the Inventory of Depressive Symptoms Self-Report (IDS-SR). A 30-item self-assessment of depressive symptoms with scores ranging from 0 (no depressive symptoms) to 90 (severe depression).
Patient Health Questionnaire 9-item | Within one week before beginning the clinical rTMS therapy course, and weekly during the clinical rTMS therapy course (typically 6 weeks), including the last day of treatment
  Scores from the Patient Health Questionnaire, 9-item version (PHQ-9). A self-assessment of depressive symptoms with scores ranging from 0 (no depressive symptoms) to 27 (severe depression).
Post-Traumatic Stress Disorder Checklist for DSM-5 | Within one week before beginning the clinical rTMS therapy course, and weekly during the clinical rTMS therapy course (typically 6 weeks), including the last day of treatment
  Scores from the Post-Traumatic Stress Disorder Checklist for DSM-5 (PCL-5). A self-assessment of PTSD symptoms with scores ranging from 0 (no PTSD symptoms) to 80 (severe PTSD symptoms)
Veteran's RAND 36-item | Within one week before beginning clinical rTMS therapy course, 3 times during the clinical rTMS therapy course (typically 6 weeks), and within one week after the conclusion of clinical rTMS therapy course
  Scores from the Veteran's RAND 36-item (VR-36). Assessment of self-reported health quality of life. Includes physical and mental component normed subscores (x=50, sd=10) ranging from 0 (worst health) to 100 (best health).

OTHER OUTCOMES:
Functional MR imaging changes related to stimulation | Within one week before beginning clinical rTMS therapy course, 3 times during the clinical rTMS therapy course (typically 6 weeks), and within one week after the conclusion of clinical rTMS therapy course
  Magnetic resonance imaging acquired throughout TMS will be analyzed to evaluate aggregate changes related to stimulation
Functional MR imaging changes predictive of outcomes | Within one week before beginning clinical rTMS therapy course, 3 times during the clinical rTMS therapy course (typically 6 weeks), and within one week after the conclusion of clinical rTMS therapy course
  Magnetic resonance imaging acquired throughout TMS will be analyzed to evaluate how brain changes can be used to predict outcomes
Functional MR imaging changes over time | Within one week before beginning clinical rTMS therapy course, 3 times during the clinical rTMS therapy course (typically 6 weeks), and within one week after the conclusion of clinical rTMS therapy course
  Magnetic resonance imaging acquired throughout TMS will be analyzed to evaluate how MR imaging of an individual changes over time

CONTACTS AND LOCATIONS:
Overall Officials: Allyson C Rosen, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA; Noah S. Philip, MD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT04016402/ICF_000.pdf